CLINICAL TRIAL: NCT06451718
Title: First in Human Study to Assess the Safety and Efficacy of an Implantable Nitinol Device in the Treatment of Stage 3 and 4 Keratoconus
Brief Title: First in Human Study to Assess Safety and Efficacy of an Implantable Nitinol Device in the Treatment of Keratoconus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recornea Srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REMKERA
Record Dates: First submitted 2024-05-07; First posted 2024-06-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Keratoconus
Keywords: GROSSO; Implant; Cornea; Surgery; Reshaper; keratoconus; keratoplasty; nitinol; corneal shape; remodeling
MeSH Terms: conditions — Keratoconus; Corneal Diseases

STUDY DESIGN:
Intervention Model Description: All enrolled subjects with keratoconus will receive the surgical intervention and will be followed for up to 1 year post-procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All participants will undergo the planned surgical intervention for the implantation of the investigational medical device and will be monitored for up to 1 year after the procedure.
  Interventions: Device: Nitinol net for intracorneal implant for keratoconus treatment

INTERVENTIONS:
Device: Nitinol net for intracorneal implant for keratoconus treatment — The investigational corneal implant device is designed for patients with keratoconus. It is intended to be surgically implanted into the cornea as a permanent implant and is made of nitinol. The device is intended to improve corneal stability and visual outcomes.

SUMMARY:
This Study is a First In Human clinical investigation addressed to evaluate the safety and efficacy of a novel intra-corneal nitinol device (Investigational Medical Device: GROSSO® implant) for the treatment of advanced keratoconus disease of the eye.

DETAILED DESCRIPTION:
The medical device under investigation is a sterile thin 8-mm diameter circular scaffold made of a nickel-titanium alloy (nitinol) that is intended as a permanent implant that is surgically inserted into the cornea in order to modify force by inducing a change in corneal shape and consequently improving vision. This study is aimed at adults with a stage 3- 4 keratoconus, a central K reading > 47.2 D and RMS of coma aberration > 2.5 μm, which are not recommended for Intrastromal Corneal Ring Segments (ICRS) and are recommended for keratoplasty. Therefore, this study represents a salvage route to preserve the cornea. Envisaged worst case scenario of failure of the experimental device patients would be redirected to keratoplasty.

Study aims to treat 12 patients separated by a safety period of at least 14 days between each one allowing safety monitoring. For each patient, the following treatment strategy will be applied:

* Unilateral KC: the affected eye meeting the eligibility criteria will be treated.
* Bilateral KC, one eye meeting the eligibility criteria: the eligible eye will be treated.
* Bilateral KC, both eyes meeting the eligibility criteria: the most severely compromised eye will be treated. Primary study objective is safety by identification or any local or systemic adverse events. Secondary objective will aim to evaluate efficacy that means a consequently improving of vision. Patients will be monitored at 1, 7, 21, 60, 180 and 365 days post implant surgery. Upon observance or any serious adverse event, increase in ocular pressure, device migration or discomfort, medical criteria or patient request, the patient will be offered for the device removed. The study will be early terminated if 3 patients have the experimental device removed for any reason or 4 patients withdraw from study.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form.
* Male and female ≥ 18 years old.
* Not recommended for ICRS.
* Recommended for keratoplasty.
* Minimum corneal thickness ≥ 350 μm.
* Best Distance Spectacle Corrected Visual Acuity (BDSCVA) with the ETDRS test ≥ 0.30 logMAR (<= 0,50 decimal notation).
* BCVA with RGP contact lens with the ETDRS test 10 letters or more than BCVA with spectacles.
* Have stable or stabilized disease for 12 months (in case of crosslinking, it must have been done at least 12 months prior to intervention).
* Have a KC stage 3-4 according to Investigator's judgement, with a central K readings > 47.2 D and RMS of coma aberration > 2.5 μm.
* Have no known or suspected allergy to nickel.
* Female subject of childbearing potential is eligible to participate if declaring she is not pregnant, or not breastfeeding and agree to use highly effective contraception (defined as method which results in a failure rate of <1% annually) and must abstain from egg donation or storage throughout the study period.

Exclusion Criteria:

* Inability of patient and/or relatives to understand the clinical investigation procedures and thus inability to give informed consent.
* Untreated progressive KC.
* Single functioning eye.
* Other ocular diseases (eyelids malposition, uveitis, ocular hypertension, glaucoma, cataract, retinal disorders) or corneal surgeries (refractive corneal surgery, keratoplasty), except corneal crosslinking.
* Systemic collagenopathies and/or vasculitis, and other diseases that in the opinion of the principal Investigator, may be contraindicated.
* Suspected or known intolerance or hypersensitivity to any of the treatments indicated in the CIP and/or to any component of the device (i.e. nickel).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Device Effects (SADE), Adverse Events (AE), and Serious Adverse Events (SAE) | From enrolment up to 12 months post-procedure
  Number and type of adverse events, serious adverse events, and serious adverse device effects observed during follow-up.
Changes in corneal alterations from baseline to 12 months. | From baseline up to 12 months post-procedure
  Slit Lamp corneal assessments to evaluate:
  * Corneal inflammation
  * Corneal infection
  * Corneal stromal lysis
  * Corneal melting
  * Corneal stromal infiltration
  * Corneal neo vessels
  * Persistent corneal epithelial defects
  Observations will be graded from 0 (Absence) to 3 (Severe)
Changes in total and epithelial corneal thickness (central and minimum) from baseline to 12 months. | From baseline up to 12 months post-procedure
  Measurement of total and epithelial corneal thickness (central and minimum)
Changes in IOP from baseline to 12 months | From baseline up to 12 months post-procedure
  IOP is measured with tonometer
Changes in corrected IOP (bIOP) from baseline to 12 months | From baseline up to 12 months post-procedure
  bIOP is measured using a biomechanically based tonometry method
Changes in macular central thickness from baseline to 12 months | From baseline up to 12 months post-procedure
  Central macular thickness is assessed with a posterior Optical Coherence Tomography (OCT).
Changes in Endothelial Cell Count (ECC) from baseline to 12 months | from baseline up to 12 months post-procedure
  Corneal endothelium assessment is performed with specular microscope
Subjective numeric scale related to several ocular symptoms | From baseline to 12 months post-procedure
  Subjective numeric scale ranked from 0 (no pain at all) to 10 (the maximum pain ever felt) related to pain, foreign body sensation, tearing, photophobia, glare and halos

SECONDARY OUTCOMES:
Changes in Best Distance Spectacle Corrected Visual Acuity (BDSCVA) from baseline to 12 months | From baseline up to 12 months post-procedure
  BDSCVA is performed using ETDRS (Early Treatment Diabetic Retinopathy Study) refraction and vision testing protocol.
Changes in topographic keratometry values from baseline to 12 months | From baseline up to 12 months post-procedure
  Corneal topography is performed by using the topographer. The values collected are Kmax, K steep, K flat and Km.
Changes in topographic and refractive astigmatism from baseline to 12 months | From baseline up to 12 months post-procedure
  Topographic astigmatism is measured in dioptres with the Topographer. Refractive astigmatism is measured in dioptres and axis, determined by refraction using ETDRS optotypes
Changes in Manifest Refraction Spherical Equivalent (MRSE) from baseline to 12 months | From baseline up to 12 months post-procedure
  MRSE is measured in dioptres, determined by refraction using ETDRS optotypes
Changes in Symmetry Index (SI) from baseline to 12 months | From baseline up to 12 months post-procedure
  SI index is measured in diopters with Topographer
Changes in Center-Surrounding Index (CSI) from baseline to 12 months | From baseline up to 12 months post-procedure
  CSI index is measured in diopters with Topographer
Assessment of the topographic centration of the implant | From surgery up to 12 months post-procedure
  Assessment of the coordinates of the centration of the device in the cornea (in dioptres and degrees).
Changes in Uncorrected Visual Acuity (UNCVA) from baseline to 12 months | From baseline up to 12 months post-procedure
  UNCVA is assessed using ETDRS
Changes in Best Corrected Visual Acuity with rigid gas permeable contact lens (RGP-BCVA) from baseline to 12 months | From baseline up to 12 months post-procedure
  RGP-BCVA is assessed in LogMAR units using ETDRS
Changes in biomechanical corneal properties expressed as Corneal Hysteresis (CH) from baseline to 12 months | From baseline up to 12 months post-procedure
  Corneal Hysteresis is measured in mmHg with the Ocular Response Analyzer (ORA)
Changes in biomechanical corneal properties, expressed as Deformation Amplitude Ratio (DA Ratio) from baseline to 12 months | From baseline up to 12 months post-procedure
  Deformation Amplitude Ratio (DA Ratio) is measured in mm/sd with Corvis ST
Changes in biomechanical corneal properties, expressed as Integrated Radius from baseline to 12 months | From baseline up to 12 months post-procedure
  Integrated Radius is measured in mm/sd with Corvis ST
Changes in biomechanical corneal properties, expressed as ARTH from baseline to 12 months | From baseline up to 12 months post-procedure
  ARTH is measured in μm/sd with Corvis ST
Changes in biomechanical corneal properties, expressed as Stiffness Parameter at first Applanation (SP-A1) from baseline to 12 months | From baseline up to 12 months post-procedure
  Stiffness Parameter at first Applanation (SP-A1) is measured in pr/mm/sd with Corvis ST
Changes in biomechanical corneal properties, expressed as Stress-Strain Index (SSI) from baseline to 12 months | From baseline up to 12 months post-procedure
  Stress-Strain Index (SSI) is calculated with Corvis ST
Changes in Vision Related Quality of Life (VRQoL) from baseline to 12 months | At screening visit (preoperatively) and at study end (12 months post-procedure)
  The NEI-42 questionnaire provides a final score reflecting vision-related quality of life. All items are scored so that higher values indicate better quality of life. Each response is converted to a 0-100 scale, where 0 represents the lowest and 100 the highest possible score. The domains evaluated include: clarity of vision, expectations, near vision, distance vision, diurnal fluctuations, activity limitations, glare, symptoms, dependence on correction, worry, suboptimal correction, appearance, and satisfaction with correction.
Stability of the corneal applanation between 6 and 12 months | Between 6 and 12 months post-procedure
  Corneal curvature or applanation is measured in dioptres, measured with a topographer
Changes in optical quality expressed as RMS from baseline to 12 months | From baseline up to 12 months post-procedure
  RMS value is measured in μm with the MS-39 topographer
Changes in optical quality expressed as OSI value from baseline to 12 months | From baseline up to 12 months post-procedure
  OSI value is measured with the HD Analizer, if available

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Grosso, MD, Study Director — Chief Medical Officer (CMO); José L. Güell, MD, Principal Investigator — Head of the Cornea, Cataract and Refractive Surgery Department at IMO
Locations (2):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Roma, Italy
- Instituto de Microcirugía Ocular de Barcelona (IMO), Barcelona, Bar, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this study will be made available upon reasonable request from qualified researchers, subject to the sponsor's discretion, in order to protect participant privacy and sponsor confidentiality.
Supporting Information: CSR

REFERENCES:
- See also: Sponsor official website — https://www.recornea.com/